CLINICAL TRIAL: NCT00700778
Title: Genomic Markers of Breast Cancer Prevention Induced by HCG in Women at High Risk
Brief Title: Recombinant Human Chorionic Gonadotropin in Preventing Breast Cancer in Premenopausal Women With BRCA1 Mutations
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit volunteers
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 06827; 06827 (Other: Fox Chase Cancer Center); R21CA124522 (NIH)
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Results first posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: BRCA1 Mutation; Breast Cancer
Keywords: breast cancer; BRCA1 mutation carrier
MeSH Terms: conditions — Breast Neoplasms | interventions — Chorionic Gonadotropin; Microarray Analysis; Immunohistochemistry; Biopsy, Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Recombinant human chorionic gonadotropin (Experimental): Patients receive recombinant human chorionic gonadotropin subcutaneously three times weekly. Treatment continues weekly for 90 days in the absence of unacceptable toxicity.
  Interventions: Biological: recombinant human chorionic gonadotropin; Genetic: microarray analysis; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Procedure: needle biopsy

INTERVENTIONS:
Biological: recombinant human chorionic gonadotropin
Genetic: microarray analysis
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Procedure: needle biopsy

SUMMARY:
RATIONALE: Chemoprevention is the use of certain drugs to keep cancer from forming. The use of recombinant human chorionic gonadotropin may prevent breast cancer in premenopausal women with BRCA1 mutations.

PURPOSE: This clinical trial is studying recombinant human chorionic gonadotropin in preventing breast cancer in premenopausal women with BRCA1 mutations.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether the genomic profiles of breast epithelial cells of high-breast cancer-risk women, as defined by their positive BRCA1 status and nulliparous condition, express a signature indicative of high-risk.

Secondary

* Determine whether women identified to express a "high-breast cancer-risk" signature will revert it to a "low-risk" signature after a 90-day treatment with r-hCG, which should have induced breast differentiation and genomic changes that would serve as biomarkers indicative of decreased breast cancer risk.

OUTLINE: Patients receive recombinant human chorionic gonadotropin subcutaneously three times weekly. Treatment continues weekly for 90 days in the absence of unacceptable toxicity.

Benign breast tissue specimens are collected by core needle biopsy at baseline, day 90, and day 270. Tissue samples are analyzed by cytopathology for epithelial normality, Ki67 immunohistochemical staining for cell proliferation, cDNA microarray for gene expression, and serum studies for hormone levels and biomarker determinations.

After completion of study treatment, patients are followed for 24 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Asymptomatic women who have a deleterious mutation on the BRCA1 gene
* Normal, no complaints, no evidence of disease
* Nulliparous, never pregnant (G0P0)
* No previous diagnosis of breast or ovarian cancer
* No known brain metastases
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* ECOG performance status (PS) 0-1 OR Karnofsky PS 90-100%
* Premenopausal with normal menstrual cycles and intact ovaries
* Normal ovarian size report from pelvic ultrasound
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to human chorionic gonadotropin preparations or one of its excipients
* No uncontrolled intercurrent illness including any of the following:

  * Ovarian enlargement of undetermined origin
  * Ovarian cysts > 2 cm
  * Microcystic ovaries, which might predispose to the development of ovarian hyperstimulation syndrome
  * History of prior cancer other than non-melanoma skin cancer
  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Severe cognitive deficit or psychiatric illness/social situations that would make her unable to give informed consent or would limit compliance with study requirements

PRIOR CONCURRENT THERAPY:

* At least 6 weeks since prior and no concurrent oral contraceptives or hormone-replacement therapy
* No concurrent tamoxifen for chemoprevention
* No concurrent participation in another chemopreventive trial for breast cancer
* No concurrent medication that could interfere with this study including any of the following:

  * Hormonal contraceptives
  * Androgens
  * Prednisone
  * Thyroid hormones
  * Insulin
* No other concurrent investigational agents
* No recent treatment with follicle-stimulating hormone for assisted reproduction
* No HIV-positive patients on concurrent combination antiretroviral therapy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2008-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jose Russo, MD, FCAP, Principal Investigator — Fox Chase Cancer Center
Locations (3):
- United States (2):
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
- Universitaetsklinik fuer Frauenheilkunde, Vienna, Austria

RESULTS

PARTICIPANT FLOW:
Groups:
- Recombinant Human Chorionic Gonadotropin: Patients receive recombinant human chorionic gonadotropin subcutaneously three times weekly. Treatment continues weekly for 90 days in the absence of unacceptable toxicity.
  recombinant human chorionic gonadotropin
  microarray analysis
  immunohistochemistry staining method
  laboratory biomarker analysis
  needle biopsy
Period: Overall Study
Arm/Group | Recombinant Human Chorionic Gonadotropin
Started | 2
Completed | 0
Not Completed | 2
Not completed — Inconclusive data due to inadequate sample collection | 2

BASELINE CHARACTERISTICS:
Population: No results were obtained
Arm/Group | Recombinant Human Chorionic Gonadotropin
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Region of Enrollment [Number; unit: participants] — No results were obtained
  participants
    Austria | 1

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Gene Expression in Breast Epithelial Cells Obtained for Asymptomatic High Breast Cancer Risk Nulliparous Premenopausal Women at Baseline, After Treatment With r-hCG at 90 Days, and at 270 Days From Baseline
Time Frame: 90 days and 270 days from baseline
Population: No results were obtained
Arm/Group | Recombinant Human Chorionic Gonadotropin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Recombinant Human Chorionic Gonadotropin
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No